CLINICAL TRIAL: NCT00653848
Title: Randomized Adjuvant Phase III Trial of Six Cycles of Docetaxel+Hormonal Treatment Versus Hormonal Treatment in Patients With Intermediate or High-risk Prostate Cancer Treated With Radical Radiotherapy
Brief Title: Adjuvant Treatment of Prostate Cancer With Docetaxel or Not After Radical Radiotherapy
Acronym: AdRad
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Scandinavian Prostate Cancer Group (Network)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPCG-13; 2006-001657-94 (EudraCT Number)
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer
Keywords: Adjuvant treatment, high risk, radical radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel arm (Experimental): six of docetaxel every third week + hormonal treatment
  Interventions: Drug: docetaxel
- Control (No Intervention): hormonal treatment only

INTERVENTIONS:
Drug: docetaxel — docetaxel 75 mg/square meter i.v. every third week, six cycles
  Other Names: LHRH ananlog 9 months
  Arms: Docetaxel arm

SUMMARY:
As docetaxel is proven to be effective in late stages of prostate cancer with a large tumour burden it should be effective in primarily treated intermediate and high risk prostate cancer as an adjuvant treatment after radiotherapy to prevent early relapse. This will therefore be tested in a randomised phase III trial where patients will be randomized either to docetaxel or surveillance

DETAILED DESCRIPTION:
Primary endpoint:

* PSA progression rate, ASTRO guidelines.

Secondary endpoints:

* PSA doubling time after progression
* Quality of Life (QoL)
* Safety
* Metastases free survival
* Overall survival

ELIGIBILITY:
Inclusion Criteria:

* Men > 18 and ≤75 years of age.
* WHO/ECOG performance status 0 - 1.
* Histological proven adenocarcinoma of the prostate within 12 months prior to randomisation
* One of the following:

  * T2 with Gleason score 7(4+3 ) and PSA >10 ng/ml to < 70 ng/ml
  * T2 with Gleason 8-10, any PSA < 70 ng/ml
  * any T3 tumour
* Prior neoadjuvant hormone therapy is mandatory for all patients
* Adequate haematological-, liver- and kidney function. (Hemoglobin > 110 g/l, neutrophils > 1.5 x 109/ l, platelets > 150 x 109/ l, ASAT and ALAT < 1.5 x ULN, ALP < 1.5 x ULN, creatinine < 1.5 x ULN)
* Written informed consent

Exclusion Criteria:

* M+
* N+ clinical or pathological
* Patients with a history of previous malignant disease. Exceptions should be made for basal cell carcinoma (BCC) and squamous cell carcinoma of the skin. Exceptions should also be made for curatively treated malignant disease, which has been disease free for the past five years.
* Previous radiotherapy to the pelvic region.
* Previous chemotherapy within 5 years.
* Systemic corticosteroids within 6 months prior to randomisation.
* Unstable cardiovascular disease, including myocardial infarction, within 6 months prior to randomisation.
* Active untreated infectious disease, including tuberculosis, MRSA.
* Active gastric ulcer.
* Known hypersensitivity to Polysorbate 80 (an excipient of docetaxel)
* Other serious illness or medical condition

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2007-05; Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
PSA progression rate | From randomization to progression
  According to RTOG-ASTRO guidelines

SECONDARY OUTCOMES:
PSA doubling time after progression, quality of life, safety, metastases free survival, overall survival | From randomisation to year 2014
  PSA doubling measured, FACT-P, detection of metastatic lesions

CONTACTS AND LOCATIONS:
Overall Officials: Pirkko-Liisa i Kellokumpu-Lehtinen, Prof, Principal Investigator — Tampere University Hospital
Locations (1):
- Jon R Iversen, Oslo, Norway